CLINICAL TRIAL: NCT03090555
Title: The Effectiveness of Translational Manipulation Under Interscalene Block for Treatment of Adhesive Capsulitis of the Shoulder: A Randomized Clinical Trial
Brief Title: Translational Manipulation Under Interscalene Block for Adhesive Capsulitis of the Shoulder (TMACS)
Acronym: TMACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel G. Rendeiro (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Daniel G. Rendeiro, Program Director, Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: c2003.176
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Shoulder Adhesive Capsulitis; Frozen Shoulder; Adhesive Capsulitis of Shoulder
Keywords: adhesive capsulitis; clinical trial; manipulation
MeSH Terms: conditions — Bursitis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are blinded to the study arm to which participants are assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Translational Manipulation (Experimental): Participants received an interscalene block on the affected side. Then, a physical therapist performed thrust manipulations on the affected shoulder until full passive physiologic motion was restored. These participants returned to the clinic approximately 3 days later for the first of 6 manual therapy (MT) sessions.
  The first clinic treatment session included instruction in a home program of static stretching, resistive exercise, and ice, issue of an illustrated handout and digital video disc detailing the same program, and manual therapy (MT) by a physical therapist that included all indicated grades of non-thrust manipulation. Subsequent clinic treatment sessions included additional MT, progression of the strengthening exercises, and reinforcement of the home program.
  Interventions: Procedure: Translational manipulation; Procedure: Manual therapy
- Comparison Group (Active Comparator): Participants in the comparison group did not undergo a session of translational manipulation. In order to equalize the number of intervention sessions, members of this group underwent 7 in-clinic sessions of manual therapy (MT). The first clinic treatment session for all study participants included instruction in the home program of static stretching, resistive exercise, and ice, issue of an illustrated handout and digital video disc detailing the same program, and MT by a physical therapist that included all indicated grades of non-thrust manipulation. Subsequent clinic treatment sessions included additional MT, progression of the strengthening exercises, and reinforcement of the home program.
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Procedure: Translational manipulation — After the patient receives an interscalene block on the affected side, a physical therapist performs a series of thrust manipulations on the participant's affected shoulder. The participant's identified limitations of physiological and accessory motion revealed during manual examination guided the physical therapist's choice of technique, which primarily consisted of an accessory superior to inferior accessory gliding motion performed in a physiological position of limited motion. Additional gliding manipulations in combined movement positions such as increased flexion or abduction plus internal or external rotation were utilized until full passive physiologic motion was restored.
  Arms: Translational Manipulation
Procedure: Manual therapy — The first clinic treatment session for all study participants included instruction in the home program of static stretching, resistive exercise, and ice, issue of an illustrated handout and digital video disc detailing the same program, and manual therapy (MT) by a physical therapist that included all indicated grades of non-thrust manipulation of the joints and soft tissue. The MT intervention was targeted toward any identifiable upper quarter pain or movement impairments. Subsequent clinic treatment sessions included additional MT, progression of the strengthening exercises, and reinforcement of the home program.

SUMMARY:
This study evaluates the addition of translational manipulation under interscalene block, to a course of orthopaedic manual physical therapy for treatment of adhesive capsulitis of the shoulder. Half the patients will receive a translational manipulation under interscalene block, plus 6 sessions of orthopaedic manual physical therapy. The other half will receive 7 sessions of physical therapy. The investigators hypothesize that the translational manipulation under interscalene block will provide additional benefit beyond the effect of in-clinic orthopaedic manual physical therapy alone.

DETAILED DESCRIPTION:
Both translational manipulation under interscalene block and in-clinic orthopaedic manual physical therapy are thought to be useful for treating adhesive capsulitis of the shoulder. However, no single intervention for this condition has been proven to be superior to others.

The translational manipulation under interscalene block may improve pain-free motion of the involved shoulder, by releasing tight tissue without the guarding and motion-limiting effect of active muscle tension. The interscalene block prevents the patient from actively contracting the muscles that control the involved shoulder, during the manipulation procedure.

One additional possible benefit of the translational manipulation under interscalene block, is that the technique loads the joint structures--bone, joint capsule--in a safer way with less angular torque than conventional/traditional manipulation under anaesthesia. This minimizes the risk of physical/mechanical harm from the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Military healthcare system beneficiaries 18 years old or older
* Chief complaint of loss of shoulder range of motion
* Passive glenohumeral abduction less than 75 degrees
* Sufficient English-language skills to understand the study protocol.

Exclusion Criteria:

* Clinical diagnosis of diabetes (type I or II)
* Clinically evident and symptomatic rotator cuff tear or cervical radiculopathy
* Pain as the primary impairment (versus limitation of motion as the primary impairment)
* Having contraindications to an interscalene block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-01-05 (Actual); Primary Completion 2006-05-31 (Actual); Study Completion 2011-04-27 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) | baseline, 3 months, 6 months, 12 months, 48 months
  Measure of individual pain and disability

SECONDARY OUTCOMES:
Percent of normal | 48 months
  Patient estimate of percent of full functional capacity of involved shoulder
Activity limitations | 48 months
  Patient estimate of identified activities limited by involved shoulder function
Medication use | 48 months
  Patient estimate of medications taken due to involved shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G. Rendeiro, DSc, Principal Investigator — Army-Baylor University Doctoral Fellowship in Orthopaedic Manual Physical Therapy
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Placzek JD, Roubal PJ, Kulig K, Pagett BT, Wiater JM. Theory and technique of translational manipulation for adhesive capsulitis. Am J Orthop (Belle Mead NJ). 2004 Apr;33(4):173-9. PMID 15132324
- [Result] Placzek JD, Roubal PJ, Freeman DC, Kulig K, Nasser S, Pagett BT. Long-term effectiveness of translational manipulation for adhesive capsulitis. Clin Orthop Relat Res. 1998 Nov;(356):181-91. doi: 10.1097/00003086-199811000-00025. PMID 9917683